CLINICAL TRIAL: NCT01023451
Title: Serum Brain Natriuretic Peptide Levels and Its Correlation With Echocardiographic Measurements Suggestive of Pulmonary Hypertension in Pediatric Patients With Sickle Cell Disease
Brief Title: Serum Brain Natriuretic Peptide Levels and Pulmonary Hypertension in Pediatric Sickle Cell Patients
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 091007
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Sickle cell disease; Pediatric patients; Brain Natriuretic Peptide levels
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is

1. To determine if Brain natriuretic peptide levels correlates with elevated tricuspid regurgitation flow velocity levels in pediatric patients with sickle cell disease
2. To determine the role of age, gender, steady state hemoglobin and disease type on Brain natriuretic peptide levels and pulmonary hypertension

DETAILED DESCRIPTION:
Pulmonary hypertension is recognized as a significant cause of morbidity and mortality in patients with sickle cell disease. Doppler echocardiography is a recommended noninvasive screening tool for sickle cell disease patients with pulmonary hypertension. Brain natriuretic peptide levels have been found to be a possible serum screening marker. This research will offer the opportunity to determine if there is any possible relationship between magnitude of BNP concentration and degree of TRV, if it can be used as a screening test in SCD pediatric patients with PHT and form the basis for a future multicenter study

ELIGIBILITY:
Inclusion Criteria:

* Male and Female any age
* Diagnosis of SCD with PHT on echocardiogram
* Controls must have a diagnosis of sickle cell disease without Pulmonary hypertension, age, gender and disease type match to subjects with pulmonary hypertension
* Parent or Legal guardian willing to sign informed consent form

Exclusion Criteria:

* Abnormal echocardiograms not related to PHT
* Parent or Legal guardian unwilling or unable to give written informed consent

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Sickle cell clinic
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Correlation of Brain Natriuretic Peptide (BNP) levels to elevated Tricuspid Regurgitation Flow Velocity (TRV) | one day
  Subjects will be asked to participate in the study by allowing a review of their echocardiographic findings. In addition, they will be asked for a 1 ml blood sample during routine annual follow ups for BNP levels to be drawn.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Do, DO, Principal Investigator — Akron Children's Hospital; Jeffrey Hord, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital Sickle Cell Clinic, Akron, Ohio, United States

REFERENCES:
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486
- [Background] Ataga KI, Sood N, De Gent G, Kelly E, Henderson AG, Jones S, Strayhorn D, Lail A, Lieff S, Orringer EP. Pulmonary hypertension in sickle cell disease. Am J Med. 2004 Nov 1;117(9):665-9. doi: 10.1016/j.amjmed.2004.03.034. PMID 15501204
- [Background] Suell MN, Bezold LI, Okcu MF, Mahoney DH Jr, Shardonofsky F, Mueller BU. Increased pulmonary artery pressures among adolescents with sickle cell disease. J Pediatr Hematol Oncol. 2005 Dec;27(12):654-8. doi: 10.1097/01.mph.0000194022.17968.bf. PMID 16344670
- [Background] Nelson SC, Adade BB, McDonough EA, Moquist KL, Hennessy JM. High prevalence of pulmonary hypertension in children with sickle cell disease. J Pediatr Hematol Oncol. 2007 May;29(5):334-7. doi: 10.1097/MPH.0b013e31805d8f32. PMID 17483714
- [Background] Castro O, Hoque M, Brown BD. Pulmonary hypertension in sickle cell disease: cardiac catheterization results and survival. Blood. 2003 Feb 15;101(4):1257-61. doi: 10.1182/blood-2002-03-0948. Epub 2002 Oct 3. PMID 12393669